CLINICAL TRIAL: NCT04892017
Title: A Phase 1/2, First-in-Human Study of DCC-3116 as Monotherapy and in Combination With RAS/MAPK Pathway Inhibitors in Patients With Advanced or Metastatic Solid Tumors With RAS/MAPK Pathway Mutations
Brief Title: A Phase 1/2 Study of Inlexisertib (DCC-3116) in Patients With RAS/MAPK Pathway Mutant Solid Tumors
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Deciphera Pharmaceuticals, LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: DCC-3116-01-001; 2022-501474-19-00 (EU CTIS Number)
Record Dates: First submitted 2021-05-06; First posted 2021-05-19 (Actual); Last update posted 2025-10-10 (Actual); Status verified 2025-10

CONDITIONS: Non-Small Cell Lung Cancer; Advanced Solid Tumor; Metastatic Solid Tumor
Keywords: KRAS G12C
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Neoplasm Metastasis | interventions — trametinib; binimetinib; sotorasib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Dose Escalation (Part 1, Cohort A Monotherapy) (Experimental): Inlexisertib tablets in escalating dose cohorts given orally twice daily (BID) in 28-day cycles as monotherapy (single agent). If no DLT in 3 participants or 1 DLT/6 participants is observed, dose escalation may continue to the next planned dose cohort.
  Interventions: Drug: Inlexisertib
- Dose Escalation (Part 1, Cohort B Combination) (Experimental): Upon determination of the RP2D/MTD single agent, inlexisertib will be dosed in combination with trametinib.
  Escalation Cohort B combination closed on January 8, 2024.
  Interventions: Drug: Inlexisertib; Drug: Trametinib
- Dose Escalation (Part 1, Cohort C Combination) (Experimental): Upon determination of the RP2D/MTD single agent, inlexisertib will be dosed in combination with binimetinib.
  Escalation Cohort C combination closed on January 8, 2024.
  Interventions: Drug: Inlexisertib; Drug: Binimetinib
- Dose Escalation (Part 1, Cohort D Combination) (Experimental): Upon determination of the RP2D/MTD single agent, inlexisertib will be dosed in combination with sotorasib.
  Interventions: Drug: Inlexisertib; Drug: Sotorasib
- Expansion Cohorts 1, 2, 3 and 4 (Part 2) (Experimental): Expansion Cohorts 1, 2, 3 and 4 inlexisertib combinations will not open for enrollment.
  Interventions: Drug: Inlexisertib
- Expansion Cohort 5 (Part 2) (Experimental): Inlexisertib tablets orally given in combination with sotorasib in 28-day cycles to evaluate safety and preliminary efficacy of participants with NSCLC (with a documented mutation in KRAS G12C).
  Interventions: Drug: Inlexisertib; Drug: Sotorasib

INTERVENTIONS:
Drug: Inlexisertib — Oral Tablet Formulation
  Other Names: DCC-3116
Drug: Trametinib — Oral Tablet Formulation
  Arms: Dose Escalation (Part 1, Cohort B Combination)
Drug: Binimetinib — Oral Tablet Formulation
  Arms: Dose Escalation (Part 1, Cohort C Combination)
Drug: Sotorasib — Oral Tablet Formulation
  Arms: Dose Escalation (Part 1, Cohort D Combination); Expansion Cohort 5 (Part 2)

SUMMARY:
This is a Phase 1/2, multicenter, open label, first in human (FIH) study of inlexisertib as monotherapy, and in combination with trametinib, binimetinib, or sotorasib in patients with advanced or metastatic solid tumors with RAS/MAPK pathway mutation. The study consists of 2 parts, a dose-escalation phase, and an expansion phase.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female participants ≥18 years of age
2. Dose Escalation Phase (Part 1):

   Escalation Cohort B combination with trametinib and Cohort C combination with binimetinib closed on January 8, 2024.
   1. Participants must have a pathologically confirmed diagnosis of an advanced or metastatic solid tumor with a documented RAS, NF1, or RAF mutations. A molecular pathology report documenting mutational status of RAS, NF1, or RAF must be available.
   2. Progressed despite standard therapies, and received at least 1 prior line of anticancer therapy.

      * Participants with a documented mutation in BRAF V600E or V600K must have received approved treatments known to provide clinical benefit prior to study entry.
   3. Participants enrolled in the inlexisertib and sotorasib cohort (Cohort D) must have a KRAS G12C mutation.
3. Dose Expansion Phase (Part 2):

   Expansion Cohorts 1, 2, 3 and 4 combinations will not open for enrollment.

   Cohort 5: Patients with KRAS G12C mutant NSCLC
   * Pathologically confirmed NSCLC with a documented mutation in KRAS G12C.
   * Received at least 1 prior line of systemic therapy in the advanced or metastatic setting.
   * Have not received prior sotorasib or other KRAS G12C inhibitor therapy.
4. Must provide a fresh tumor biopsy from a primary or metastatic cancer lesion if it can be biopsied with acceptable risk as determined by the Investigator.
5. Must have at least 1 measurable lesion according to Response Evaluation Criteria in Solid Tumors (RECIST), v1.1
6. Eastern Cooperative Oncology Group (ECOG) score of 0 to 2 (Dose Escalation) or 0 to 1 (Dose Expansion) at Screening
7. Adequate organ function and bone marrow function.
8. If a female of childbearing potential must have a negative pregnancy test prior to enrollment and agree to follow the contraception requirements.
9. Male participants must agree to follow contraception requirements.
10. Must provide signed consent to participate in the study and is willing to comply with study-specific procedures.

Exclusion Criteria:

1. Must not have received the following within the specified time periods prior to the first dose of study drug:

   1. Prior therapies (anticancer or therapies given for other reasons) that are known strong or moderate inhibitors or inducers of CYP3A4 or P-glycoprotein (P-gp) including certain herbal medications (e.g., St. John's Wort): 14 days or 5× the half-life of the medication (whichever is longer)
   2. All other prior anticancer therapies or any therapy that is investigational for the participant's condition with a known safety and PK profile: 14 days or 5× the half-life of the medication (whichever is shorter)
   3. Investigational therapies with unknown safety and PK profile: 28 days. If there is enough data on the investigational therapy to assess the risk for drug-drug interactions and late toxicities of prior therapy as low, the Sponsor's Medical Monitor may approve a shorter washout of 14 days
   4. Grapefruit or grapefruit juice: 14 days
2. Has a prior or concurrent malignancy that requires treatment or is expected to require treatment for active cancer during this study . Hormonal maintenance after treatment is allowed.
3. Have not recovered from all toxicities from prior therapy according to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE).
4. Presence or history of central nervous system (CNS) metastases or leptomeningeal disease, with some exceptions
5. New York Heart Association Class III or IV heart disease, active ischemia, or any other uncontrolled cardiac condition such as angina pectoris, clinically significant cardiac arrhythmia requiring therapy, uncontrolled hypertension, congestive heart failure, or myocardial infarction within 6 months prior to the first dose of study drug.
6. Prolongation of the QT interval corrected by Fridericia's formula (QTcF) based on repeated demonstration of QTcF >450 ms in males or >470 ms in females at screening, or history of long QT syndrome.
7. Left ventricular ejection fraction (LVEF) <50% at Screening
8. Systemic arterial thrombotic or embolic events within 6 months prior to the first dose of study drug
9. Systemic venous thrombotic events within 1 month prior to the first dose of study drug
10. Malabsorption syndrome
11. Major surgery within 4 weeks of the first dose of study drug. All surgical wounds must be healed and free of infection or dehiscence before the first dose of the study drug.
12. Any other clinically significant comorbidities.
13. For participants receiving inlexisertib and trametinib combination or inlexisertib and binimetinib combination: previous treatment with trametinib or binimetinib that resulted in treatment discontinuation due to intolerability as a result of an adverse event (AE) that was considered related to trametinib or binimetinib.
14. For participants receiving inlexisertib and sotorasib combination in Dose Escalation Part 1: previous treatment with sotorasib that resulted in treatment discontinuation due to intolerability as a result of an adverse event (AE) that was considered related to sotorasib.
15. For participants receiving inlexisertib and sotorasib combination: Use of proton pump inhibitors (PPIs) and H2 receptor antagonists that cannot be discontinued 3 days prior to the start of study drug administration.
16. Known allergy or hypersensitivity to any component of the investigational drug products.
17. Known human immunodeficiency virus unless the following requirements are met:

    1. CD4 count >350/µL
    2. No AIDS-defining opportunistic infection in the last 12 months
    3. Stable anti-retroviral regimen with medications that are not prohibited by the protocol for at least 4 weeks with HIV viral load less than 400 copies/mL prior to enrollment.
18. Known active hepatitis B, active hepatitis C infection or if the participant is taking medications that are prohibited per protocol.
19. If female, the participant is pregnant or lactating.
20. Ongoing participation in an interventional study.
21. For participants receiving inlexisertib and binimetinib combination: Known Gilbert's syndrome

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Estimated)
Dates: Start 2021-06-15 (Actual); Primary Completion 2027-08 (Estimated); Study Completion 2028-08 (Estimated)

PRIMARY OUTCOMES:
Incidence of Adverse Events | Approximately 24 months
  Identify the observed adverse events, serious adverse events associated with inlexisertib as monotherapy and in combination with trametinib, binimetinib, or sotorasib.
Maximum tolerated dose (MTD) (Escalation Phase) | Approximately 18 months
  Identify the dose-limiting toxicities for each dose level tested and determine the maximum tolerated dose/recommended Phase 2 doses of inlexisertib as monotherapy and in combination with trametinib, binimetinib, or sotorasib.
Objective response rate (ORR) (Expansion Phase) | Approximately 24 months
  Proportion of participants who achieve CR or PR per RECIST v1.1.

SECONDARY OUTCOMES:
Duration of response (DoR) | Approximately 24 months
  DoR is defined as the time interval from the time that the measurement criteria are first met for CR or PR (whichever is first recorded) until the first date that the progressive disease is objectively documented or death, whichever occurs first.
Disease Control Rate (DCR) | Approximately 24 months
  The DCR is defined as the proportion of participants who achieve CR, PR, or stable disease (SD) at the specified time point per RECIST v1.1.
Time to response | Approximately 24 months
  Time to response is defined as the time from initiation of treatment until the first assessment demonstrating CR or PR per RECIST v1.1.
Progression-free survival (PFS) | Approximately 24 months
  PFS is defined as the time from initiation of treatment until documented disease progression per RECIST v1.1 or death, whichever occurs first.
Maximum observed concentration (Cmax) | Predose and up to 12 hours postdose
  Measure the maximum observed concentration of inlexisertib (single-agent and combinations).
Time to maximum observed concentration (Tmax) | Predose and up to 12 hours postdose
  Measure the time to maximum plasma concentration of inlexisertib (single-agent and combinations).
Minimum observed concentration (Cmin) | Predose and up to 12 hours postdose
  Measure the minimum observed concentration of inlexisertib (single-agent and combinations).
Area under the concentration-time curve (AUC) | Predose and up to 12 hours postdose
  Measure the AUC of inlexisertib (single-agent and combinations).

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Team, Study Director — Deciphera Pharmaceuticals, LLC
Locations (10):
- United States (10):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Washington University Siteman Cancer Center, St Louis, Missouri
  - Rutgers Cancer Institute, New Brunswick, New Jersey
  - Laura & Isaac Perlmutter Cancer Center at NYU Langone Health, New York, New York
  - Oregon Health and Science University, Portland, Oregon
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - NEXT Oncology, Austin, Texas
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
  - NEXT Oncology, San Antonio, Texas
  - University of Wisconsin Clinical Science Center, Madison, Wisconsin